CLINICAL TRIAL: NCT04394221
Title: Oral Health Related Quality of Life and Parental Perception in A Group of Children and Adolescents With Down Syndrome: A Cross-Sectional Study
Brief Title: OHRQoL and Parental Perception in a Group of Children and Adolescents With Down Syndrome: A Cross
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Ahmed Essam Ahmed Ali, principal investigator Amr Ahmed Essam Ahmed, Cairo University
Other Study IDs: OHRQoL in down syndrome
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Quality of Life; Down Syndrome; Oral Health
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate Oral Health related quality of life of children and adolescents with down syndrome and Parental Perception, knowledge and Attitude on oral health conditions of children and adolescents with down syndrome

DETAILED DESCRIPTION:
Oral disease and conditions can undermine self-image and self-esteem , dis-courage normal social interaction, and cause other health problems and lead to chronic stress and depression , They may also interfere with vital-functions such as breathing , food selection eating, swallowing and speaking, and with activities of daily living such as work, school, and family interactions .

Oral Health Related Quality of Life captures the aim of new prospective and defined as a multidimensional construct that reflects people's comfort when eating, sleeping and engaging in social inter-action, their self-esteem and their satisfaction with respect to their oral health .

Down syndrome (DS) is the most common neuro-developmental disorder of known genetic origin, arising from an extra copy of chromosome 21.

Children and adolescents with down syndrome present particular characteristics that may have a negative impact on their oral health and function. Protruding large tongue and facial muscle hypotonicity impairing speaking and chewing abilities. Bruxism, respiratory problems and mouth breathing are common among them.

Periodontal disease is the most significant oral health problem in people with Down syndrome due immunological deficiency, poor masticatory function and poor oral hygiene .

Another common oral manifestation associated with the syndrome is malocclusion. In this regard, mandibular protrusion, anterior open bite, and posterior crossbite have been reported as prevalent outcomes among DS individuals .

It has been shown that the impact of oral disease on Oral Health Related Quality Of Life of children with disabilities can be used in health service planning and priority setting.

Studies have recommended that people with a negative oral condition should receive treatment first , Hence this vulnerable group of children needs to be prioritized in the planning of health services and oral health care programs

ELIGIBILITY:
Inclusion Criteria:

* Parents of children and adolescents diagnosed with Down syndrome who agree to participate in the study.
* Children and adolescents with Down syndrome aged from 4 to 14 years.
* Both genders.

Exclusion Criteria:

-Children/adolescents with multiple disabilities

Ages: 4 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Children and adolescents with down syndrome present particular characteristics that may have a negative impact on their oral health and function such as Protruding large tongue , facial muscle hypotonicity impairing speaking and chewing abilities,bruxism, respiratory problems and mouth breathing are common among them ,Periodontal disease is the most significant oral health problem in people with Down syndrome due immunological deficiency, poor masticatory function and poor oral hygiene
Sampling Method: Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
oral health related quality of life of children with down syndrome | one week
  oral health related quality of life of children with down syndrome will be measured by using Brazilian version of the Oral Health Scale for People with Down syndrome by using scoring system Scoring system Not at all =0 A little=1 Quite a lot =2 Very much =3 the minimum value is 0 the maximum value is 3 and higher scores mean a worse outcome

SECONDARY OUTCOMES:
Parental perception (knowledge and Attitude on oral health conditions) of children and adolescents with Down syndrome | one week
  Parental perception (knowledge and Attitude on oral health conditions) of children and adolescents with Down syndrome will be mesured and known by using Brazilian version of the Oral Health Scale for People with Down syndrome by using scoring system Scoring system Not at all =0 A little=1 Quite a lot =2 Very much =3 the minimum value is 0 the maximum value is 3 and higher scores mean a worse outcome in addition to using mcq questions from oral health questionnaire for parental knowledge and Attitude on their children oral health with down syndrome by using simple MCQ questions and the results will be presented in percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Facult, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bennadi D, Reddy CV. Oral health related quality of life. J Int Soc Prev Community Dent. 2013 Jan;3(1):1-6. doi: 10.4103/2231-0762.115700. PMID 24478972
- [Background] Satcher D, Nottingham JH. Revisiting Oral Health in America: A Report of the Surgeon General. Am J Public Health. 2017 May;107(S1):S32-S33. doi: 10.2105/AJPH.2017.303687. No abstract available. PMID 28661821
- [Background] Karmiloff-Smith A, Al-Janabi T, D'Souza H, Groet J, Massand E, Mok K, Startin C, Fisher E, Hardy J, Nizetic D, Tybulewicz V, Strydom A. The importance of understanding individual differences in Down syndrome. F1000Res. 2016 Mar 23;5:F1000 Faculty Rev-389. doi: 10.12688/f1000research.7506.1. eCollection 2016. PMID 27019699
- [Background] Hennequin M, Faulks D, Veyrune JL, Bourdiol P. Significance of oral health in persons with Down syndrome: a literature review. Dev Med Child Neurol. 1999 Apr;41(4):275-83. doi: 10.1017/s0012162299000596. No abstract available. PMID 10355815
- [Background] Kaye PL, Fiske J, Bower EJ, Newton JT, Fenlon M. Views and experiences of parents and siblings of adults with Down Syndrome regarding oral healthcare: a qualitative and quantitative study. Br Dent J. 2005 May 14;198(9):571-8, discussion 559. doi: 10.1038/sj.bdj.4812305. PMID 15895058
- [Background] Allen PF. Assessment of oral health related quality of life. Health Qual Life Outcomes. 2003 Sep 8;1:40. doi: 10.1186/1477-7525-1-40. PMID 14514355
- [Background] Glassman P, Miller CE. Effect of preventive dentistry training program for caregivers in community facilities on caregiver and client behavior and client oral hygiene. N Y State Dent J. 2006 Mar-Apr;72(2):38-46. PMID 16711592
- [Background] Norwood KW Jr, Slayton RL; Council on Children With Disabilities; Section on Oral Health. Oral health care for children with developmental disabilities. Pediatrics. 2013 Mar;131(3):614-9. doi: 10.1542/peds.2012-3650. Epub 2013 Feb 25. PMID 23439896
- [Background] Porovic S, Zukanovic A, Juric H, Dinarevic SM. ORAL HEALTH OF DOWN SYNDROME CHILDREN IN BOSNIA AND HERZEGOVINA. Mater Sociomed. 2016 Oct;28(5):370-372. doi: 10.5455/msm.2016.28.370-372. Epub 2016 Oct 17. PMID 27999487